CLINICAL TRIAL: NCT05845255
Title: Clinical Study for the Validation of the Medical Device Mjn-SERAS for the Detection and Prediction of Epileptic Seizures in Individuals from 12 to 65 Years, Suffering from Drug-resistant Epilepsy During Their Day-to-day Activity, to Find Out the Impact of the Digital Solution in the Quality of Life in a Normalised Environment and Provide Valuable Information from Real-World Data.
Brief Title: Evaluation of the Epilepsy-related Quality of Life, Seizure-related Accidents and Validation of the Mjn-SERAS Solution in the Normalised Patient Environment with Real-World Data
Acronym: SERAS_Home_RWD
Status: Recruiting | Type: Observational
Sponsor: MJN Neuroserveis, S.L (Industry)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Oxford University Hospitals NHS Trust (Other); Diakonie Kork (Unknown); Clínica Corachan (Unknown)
Responsible Party: Sponsor
Other Study IDs: 04_SERAS_Home_RWD
Record Dates: First submitted 2023-03-21; First posted 2023-05-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Quality of Life; Epilepsy (treatment Refractory)
Keywords: Safety and Performance; Medical device; Quality of life
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: mjn-SERAS — Using of wearable, non-invasive device for EEG recording and forecasting of epileptic seizures

SUMMARY:
The study will be prospective, multicentre, postmarketing clinical study, with a controlled and randomized design, to perform the analysis of 130 subjects with a clinical diagnosis of epilepsy, patients whose clinical semiology of their epilepsy is considered to be of interest for the validation in the day-to-day life a medical device (mjn-SERAS), which has already been validated and certified in Europe with CE mark Class IIa.

This new validation will take place in the participant's normalised environment, in individuals between 12 and 65 years of age, of both sexes with a diagnosis of drug-resistant epilepsy to determine the impact in quality of life of the mjn-SERAS on the early detection of epileptic seizures and the generation of a pre-seizure alert with a time window of a minimum of 1 minute.

DETAILED DESCRIPTION:
A prospective, multicentre, postmarketing, with a controlled and randomized design, clinical study is proposed to validate in the day-to-day life a medical device (mjn-SERAS), which has already been validated and certified in Europe by BSI(British Standard Institution) Group (CE2797) notified body CE 685187. The study will be performed in Spain, Germany and UK (United Kingdom).

The patient's characteristics about epilepsy, drug-resistant epilepsy, inclusion and exclusion criteria for the study, considering the same classification in ICD-10 (International Statistical Classification of Diseases) for Spain and NHS(National Health Services) in the UK, and ICD(International Classification of Diseases) ICD-10-GM for Germany, and the target population where the researchers will study the solution are the same for the 3 countries, so all are considering the international standards from ILAE(International League Against Epilepsy) 2017 classification, including German Society for Epileptology and ILAE British Chapter, defined in next sections.

This new validation will take place in the participant's normalised environment, in individuals between 12 and 65 years of age, of both sexes with a diagnosis of drug-resistant epilepsy, according to CE mark considerations and intended use, which will make it possible to determine the impact of the mjn-SERAS on the early detection of epileptic seizures and the generation of a pre-seizure alert with a time window of a minimum of 1 minute. The sensitivity, specificity and accuracy of the medical device solution in the studied environment will also be calculated.

The pre-determined sample size determined is an n=130 exposed individuals who meet the inclusion criteria. The patients will be recruited in Spain, Germany, and UK. The pre-post assessment for each patient will allow to compare data before and after the use of the mjn-SERAS solution, creating a baseline initially and a final evaluation. A control group will be randomized to assess the difference between both groups.

The method applied during the study consists of using a mjn-SERAS, software application with the earpiece of the external auditory canal customised for the patient.

From a methodological point of view, the general clinical variables to be included are the number of seizures (determining the onset of the seizure according to medical criteria), the type of seizure, semiological characteristics, duration, identification of the lateralisation of the epileptic focus, type of epilepsy, aetiology and pharmacological resistance. The patient will also be asked to report all the alarms and seizures using a simple app on his/her mobile phone in order to subsequently analyse and determine the results according to the patient's own experience.

Chronologically the study will be split in 3 phases and 4 periods:

* Phase 1, Baseline

  * T0 period, 2 months after recruiting for baseline creation, questionnaires, and quality of life.
* Phase 2, Intervention

  * T1 period, 4 to 10 weeks minimum, for artificial intelligence algorithm training with real seizures from the patients.
  * T2 period, 6 months minimum, for run-time algorithm, seizure risk alert mode.
* Phase 3, Results

  * T3 period for closing and comparing with baseline, questionnaires, and quality of life.

The improvement in quality of life will be assessed in a Randomized Control Trial design plus a pre-post assessment, comparing the initial questionnaires from T0 period with the ending questionnaires from T3 period. There will be several questionnaires, epilepsy specific questionnaire for Quality of Life as QOLIE-31, and generic as EQ-5D-5L. Also, questionnaires as HADS, SCL-90-R and PAM-13 will be performed for anxiety, depression, hostility, physical functioning and role limitations dimension.

The digital solution is composed by a software application in the mobile phone and a recording wearable. The application is based on artificial intelligence algorithms to generate the alerts and warning for the patient, receiving a visual, vibration and sound alert when the level is reaching the high risk, allowing the patient to take personal safety measures, that are not included in the protocol.

The main functionalities are the warning system, the calendar of seizures and the information for the patient.

The main functionalities of mjn-SERAS solution are applied to improve the quality of life of patients and improve their safety regarding epilepsy seizures. Receiving seizure alerts before they happen implies a great advantage for these patients, since the main problem with epileptic seizures is the uncertainty of when the next seizure will be, which generates a state of anxiety and constant vigilance, both for the patients and for their relatives.

Receiving an alert, a notice, before the seizure will allow them to be safe and avoid accidents and injuries caused by the seizure, which will still happen, but with less impact on the person. Just being able to reduce the state of anxiety of the person represents a very considerable improvement in the quality of life, medical benefit, since the stress indices will drop, and the person's safety will rise. Therefore, we can allow the person to carry out certain activities that until now were limited, such as walks, shopping, better schooling, social activities, so that their autonomy is greatly increased.

This increase in autonomy is closely related to the possibility of avoiding accidents and injuries caused by seizures, so that by suffering the seizure in a more controlled environment we can avoid many negative consequences and increase the patient safety.

Avoiding accidents, improving the quality of life and improving social relationships makes the person have an improvement in their state of health, since they will have fewer injuries and fewer side effects due to these seizures.

The patient will have a digital diary of the seizures to report date and time of the seizure, as well as other information, intensity of the seizure(duration) and accidents caused by the seizure.

The reports may include both real seizures and those detected by the patients, as well as two other types: psychogenic seizures that patients suffer but do not have an electrical manifestation on the EEG and, on the other hand, subclinical seizures, with an electrical manifestation on the EEG but without clinical manifestation in the patient.

All these data will be extracted from the application in an easy way, with a friendly interface according to specific guidelines, with a printable form and human-readable information. It is a pdf document that the patient can easily download and share with medical professionals.

The Epilepsy management service, is an educational feature that will help patients in their day-to-day life, it is composed by useful information containing for each country and language:

* Information about the disease
* Classification of seizures
* Epilepsy treatments and medications
* What to do in a seizure
* Links of interest

  * Patients' associations in their country
  * Regional societies of epilepsy
  * Clinical centers
  * Useful information in videos It is a dynamic information based on a webview connection in the application, where information is updated periodically and with the possibility of adding features online without necessity of update in the patient application.

ELIGIBILITY:
Inclusion Criteria:

* Age criterion:

  o Patient must be 12 to 65 years of age inclusive, at the time of signing the informed consent.
* Clinical criteria:

  * Confirmed diagnosis of drug-resistant*1 epilepsy, with focal, generalized or focal -generalized seizures, according to international standards from ILAE 2017 classification*2 (link), who will be evaluated by a specialised epilepsy unit and who are expected to have seizures.
  * The video-EEG records of patients must have epileptic seizures counted and recorded by specialised clinical personnel through accepted and contrasted gold-standard systems*3 or evaluated by a specialized epilepsy unit and expected to experience seizures with electroclinical manifestations If there are clear clinical epileptic seizures (e.g. motor seizures), patients could be involved even without v-EEG records, according to medical criteria.
  * Patients with a clinical history and previous video-EEG records that allows certainty about the diagnosis and characteristics of the participant's epilepsy. If there are clear clinical epileptic seizures (e.g. motor seizures), patients could be involved even without v-EEG records, according to medical criteria.
  * Precise semiological information on the patients included.
  * Patients with both sides localisation will be accepted, and the wearable device will be placed in the side that is most evident the origin of the seizures, to be placed as near as possible to the focal point.
  * Presence of more than 10 day seizures per year, from tonic, tonic-clonic, clonic or atonic seizures, and a minimum of 2 to 4 day seizures per month (preferably 4 per month/ 1 per week) during the last 3 months, reported by the patients/caregivers or assessed by the neurologist through the patient history. The patient must have seizures during the day to record them, not just seizures at night.
  * Patients included in ICD-10*4 and ICD-10-GM*5 classification as G40 with electroclinical manifestation of seizures.
* G40.1 Localization-related (focal) (partial) symptomatic epilepsy and epileptic syndromes with simple focal seizures
* G40.2 Localization-related (focal) (partial) symptomatic epilepsy and epileptic syndromes with complex focal seizures
* G40.3 Generalized idiopathic epilepsy and epileptic syndromes
* G40.6 Grand mal seizures, unspecified (with or without petit mal). According to medical criteria and electroclinical seizure manifestations (focal, focal-generalized or generalized onset seizure with a normal interictal EEG recording).
* G40.8 Other epilepsies (Epilepsies and epileptic syndromes, undetermined whether focal or generalized). According to medical criteria and electroclinical seizure manifestations (focal, focal-generalized or generalized onset seizure with a normal interictal EEG recording).

  o In case of epileptic syndromes not listed in the above or shows some of the syndromes mentioned in the exclusion criteria, patients could be included according to medical criteria defined by the clinician. These criteria must be accordingly justified by the clinician ( e.g., focal or generalized onset seizures without encephalopathy and with a normal interictal EEG recording).
* Technological criteria:

  * Ability to navigate in Android or iOS operating system. If mild or moderate disability, family members can assist with navigation if patient is unable. The smartphone must stays with the patient to record EEG, but seizures are registered by a family member.

Exclusion criteria

* Presence of psychogenic seizures.

  * If there is a coexistence of epileptic and non-epileptic seizures, it will be considered an exclusion criterion if the patient or family cannot differentiate between the two types of seizures.
  * If the patient or family can always differentiate between the two types of seizures, the patient could be included in the study according to medical criteria (but only recording the epileptic seizures.)
* Psychiatric, neurological, or systemic disorders that the researcher believes could affect the realisation and interpretation of the results.
* Presence of more than 10 seizures per day on a habitual basis.
* Presence of epilepsia partialis continua (G40.5*4*5)
* Patients with legal representative
* Pregnant women
* Patients with only absence seizures (G40.A*4,G40.4*5)
* Patients with only myoclonic seizures or epileptic spasms (G40.B*4,G40.4*5).
* Patients included in ICD-10*4 and ICD-10-GM*5 classification and not included in the medical criteria for specific epileptic syndromes in inclusion criteria.

  * G40.0 Localization-related (focal)(partial) idiopathic epilepsy and epileptic syndromes with seizures of localized onset
  * G40.4 Other generalized epilepsy and epileptic syndromes. In case of specific epileptic syndromes, patients could be included according to medical criteria (e.g., focal or generalized onset seizures without encephalopathy and with a normal interictal EEG recording)
  * G40.5 Epileptic seizures due to external causes*4 or Special epileptic syndromes*5
  * G40.7 Petit mal, unspecified, without grand mal seizures
  * G40.9 Epilepsy, unspecified
* Participants in previous clinical trials with mjn-SERAS device.
* In the case the patient presents an epileptic syndrome mentioned in the exclusion criteria, the patient if the clinician considers the subject meets medical criteria to be included, the patient can be enrolled in the study. These criteria must be accordingly justified by the clinician (e.g., focal or generalized onset seizures without encephalopathy and with a normal interictal EEG recording

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to the 2005 World Health Organization (WHO) report, epilepsy is a disease that affects about 1% of the population worldwide. 30% of patients are resistant to antiepileptic treatment.
  It is proposed a clinical trial for people from 12 to 65 years, in a day-to-day activity outside hospital. It will be a prospective analysis of 130 subjects with a clinical diagnosis of epilepsy patients whose clinical semiology of their epilepsy is considered to be of interest for the validation of this study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life index of patients with epilepsy | 6 months
  1. To assess the quality of life of patients with epilepsy and the degree of health perceived by the patient when using the mjn-SERAS solution to generate alarms when the possibility of a new epileptic seizure is anticipated.
  • Endpoint : Change from baseline in the epilepsy-related quality of life (QOLIE-31 questionnaire for adults 18 to 65 and QOLIE-AD-48 questionnaire for adolescents 12 to 17) after the use of the mjn-SERAS solution during T2 period, assessed in T3 period and including pre-post assessment and comparison between intervention and control group.
  • Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period) QOLIE-31, Quality of Life Index Epilepsy and QOLIE-AD-48
Patient's safety associated with seizure-related accidents | 6 months
  2. To assess the evolution of the patient's safety related with seizure-related accidents in patients with epilepsy when using the mjn-SERAS solution.
  * Endpoint Change from baseline in the number of seizure-related accidents and injuries during the use of the mjn-SERAS solution in the T2 period, assessed in T3 period, including pre-post assessment and comparison between intervention and control group.
  * Evaluation Evaluation will be performed at the T3 period with a comparison of number and severity of accidents between control group, as baseline, and intervention group, using the device.

SECONDARY OUTCOMES:
Change in health resources utilization | 12 months
  5. Assess the impact on health care resources utilization (including associated sick leave) as a result of the ability to take preventive measures ahead of a seizure.
  * Endpoint :
    o Change in use of healthcare resources, variation in frequency of use of resources, for mjn-SERAS solution, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation :
    * Healthcare resources*1 related to seizures during at least 2 months before and after starting to use the mjn-SERAS will be collected.
    * Days of sick leave due to seizures (only in patients actively employed) and hours per week needing a caregiver (informal care) in each period will also be collected.
  Healthcare resources*1: Health care resources related to seizures are number of visits to general practitioner, specialists and emergency room, hospitalizations, outpatient procedures, hours of formal care and unscheduled visits or any other use of resources.
Seizure correlation for patients report | 12 months
  6a. Measure the correlation between the warning alarms of mjn-SERAS solution and the report provided by the patient/caregiver/families regarding the presence of clinically significant epileptic seizures, as well as to analyse the algorithm for evaluating the possibility of seizure presentation and its subsequent correlation and agreement with the clinical phase.
  * Endpoints :
    * Correlation of seizures with patient report and the reliability of mjn-SERAS reports for the coordination of treatment processes with healthcare providers at T3 period, end of T2 period, 6 months minimum.
  * Evaluation :
  * The report provided by patients/caregiver is assumed as the criterion for the presence of seizures, validated by a double check, automatic seizure detection soft, automatic review, and neurologist review, human review.
Change in quality of life 5D of patients with epilepsy | 6 months
  1. To assess the quality of life of patients with epilepsy and the degree of health perceived by the patient and caregiver when using the mjn-SERAS solution to generate alarms when the possibility of a new epileptic seizure is anticipated.
  * Endpoints :
    o Change in the health-related quality of life (EQ-5D-5L) after the use of the mjn-SERAS solution at T3 period, end of T2 period, 6 months minimum.
  * Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period) o EQ-5D-5L
Change in social relationships and role limitations | 12 months
  4. To analyse the evolution of social relationships indicators in different areas of personal development in patients with epilepsy who regularly use the MJN SERAS solution.
  * Endpoints :
    o Change in role limitations due to physical health (SF-36) and autonomy of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period) o Role limitations due to physical health in SF-36.
Change in mental and emotional well-being | 12 months
  3. To analyse the change in the mental and emotional well-being of patients with epilepsy who regularly use the mjn-SERAS solution.
  * Endpoints :
    * Change in emotional well-being and quality of life (SCL-90-R Anxiety dimension) of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum.
    * Change in emotional well-being and quality of life (SCL-90-R Depression dimension) of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum.
    * Change in emotional well-being and quality of life (SCL-90-R Hostility dimension) of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period)
    * Questionnaire SCL-90-R Anxiety dimension.
    * Questionnaire SCL-90-R Depression dimension.
    * Questionnaire SCL-90-R Hostility dimension.
Seizure correlation for patient knowledge | 12 months
  6b. Measure the correlation between the warning alarms of mjn-SERAS solution and the report provided by the patient/caregiver/families, as well as to analyse the algorithm for evaluating the possibility of seizure presentation and its subsequent correlation and agreement with the clinical phase.
  * Endpoints :
    o Change in the communication between patients and healthcare providers, and the coordination of treatment processes, adapting the therapy to the real needs of the patient, with a Patient Knowledge questionnaire, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation :
    * Creation of a baseline in the Patient knowledge questionnaire (link) with questions to doctors and KOL(Key Opinion Leaders), asking for the expectations about the use of similar solutions and performing a post-assessment with the clinical professionals involved in the study about the accomplishment of these expectations. (Pre-Post assessment)
Medical device performance | 12 months
  7. To analyse and validate the mjn-SERAS solution in the standard patient environment as a system for assessing the possibility of epileptic seizures, generating an alarm prior to the clinical evidence or manifestation of a seizure to avoid accidents*2
  * Endpoint :
    o mjn-SERAS medical device performance*3 at the end of T2 period, 6 months minimum.
  * Evaluation : percentage rates of the digital solution
    * Sensitivity (rate of assessment of positive seizure possibilities with a positive clinical episode)
    * Specificity (rate of assessment of a negative seizure possibility with a negative clinical episode)
    * Accuracy (positive predictive value, PPV)
    * F-Score (weighted average of accuracy, accuracy, considering the imbalance of cases)
  Medical device performance*3: "Performance of a clinical function, other than that related to basic safety, where loss or degradation beyond the limits specified by the manufacturer results in an unacceptable risk."
Device safety evaluation with questionnaire | 12 months
  8. To analyse the usability and device-related safety of the digital solution in normal life conditions, normalised environment, with a daily use by the patient.
  * Endpoint :
    * Device safety evaluation, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation :
    * Study questionnaire, Device dimension (Post assessment) (Questionnaires definition link)
Device safety evaluation and adverse effects | 12 months
  8. To analyse the usability and device-related safety of the digital solution in normal life conditions, normalised environment, with a daily use by the patient.
  * Endpoint :
    * Device safety evaluation, at T3 period, end of T2 period, 6 months minimum.
  * Evaluation :
    * Adverse effects notification, Clinical Investigational Report (CIR)

OTHER OUTCOMES:
Specification of patients for the use of mjn-SERAS solution | 12 months
  9. The creation of a database that allows the relation of semiological variables, location of the epileptic focus and the specific results of the mjn-SERAS solution in each of the cases.
  * Endpoint :
    * Specification of patients for the use of the mjn-SERAS solution
  * Measurement :
    * Segmentation of the cases through artificial intelligence using as features the EEG parameters and the clinical variables
Specification of seizures for AI(Artificial Intelligence) algorithm | 12 months
  10. To analyse the results of the mjn-SERAS solution according to the different crisis semiology.
  * Endpoint :
    * Specification of seizures for artificial intelligence algorithm
  * Measurement : Segmentation of different semiologies to compare the ratios
    * TPR(sensitivity, True Positive Rate)
    * TNR(specificity, True Negative Rate)
    * PPV(Positive Prediction Value)
    * FAR(False Alarm Rate)
Knowledge dissemination to doctors | 12 months
  11. To increase the knowledge of healthcare professionals on the patient and the disease, by way of accessing EEG records and seizures to make better decisions on treatment and therapies .
  * Endpoint :
    * Knowledge dissemination to doctors and scientific community
  * Evaluation :
    * Creation of a baseline with questions to physicians about patient knowledge in seizures and medication, as well as performing a post-assessment with the clinical professionals involved in the study. (Pre-Post assessment)
Change in social relationships and physical functioning | 12 months
  4. To analyse the evolution of social relationships indicators in different areas of personal development in patients with epilepsy who regularly use the MJN SERAS solution.
  * Endpoints :
    o Change in physical functioning dimension (SF-36) of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum
  * Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period) o Physical functioning dimension in SF-36.
Change in quality of life social relationships | 12 months
  4. To analyse the evolution of social relationships indicators in different areas of personal development in patients with epilepsy who regularly use the MJN SERAS solution.
  * Endpoints :
    o Change in social relationships dimension (QOLIE-31) of the patient after the use of the mjn-SERAS, at T3 period, end of T2 period, 6 months minimum
  * Evaluation : Questionnaires answered by patients (Pre-Post assessment, baseline vs T3 period) o Social relationships dimension in QOLIE-31.
Knowledge dissemination to scientific community | 12 months
  11. To increase the knowledge of healthcare professionals on the patient and the disease, by way of accessing EEG records and seizures to make better decisions on treatment and therapies .
  * Endpoint :
    * Knowledge dissemination to doctors and scientific community
  * Evaluation :
    * Reports and publications

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Nagel, MD PhD, Principal Investigator — Department of Neuroscience Clinica Corachan & Synaptia Health Projects
Locations (6):
- Diakonie Kork, Kork, Germany
- Spain (4):
  - Clínica Corachan, Barcelona, Barcelona
  - CUN, Madrid, Madrid
  - Vithas La Milagrosa, Madrid, Madrid
  - CUN, Pamplona, Navarre
- Oxford NHS, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided